CLINICAL TRIAL: NCT01668420
Title: Effect of Thermal Stimulation for Lower Extremity Movement and Function in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hsin-Wen Hsu (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Hsin-Wen Hsu, physical therapist (graduated student), Kaohsiung Medical University Chung-Ho Memorial Hospital
Organization: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMUH-IRB-980332
Record Dates: First submitted 2012-08-12; First posted 2012-08-20 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: thermal stimulation; lower extremity; temperature; efficacy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- noxious thermal stimulation (Experimental): Heat-pain:46-47°C and Cold-pain:2-3°C alternately (intervention) 3 times /week and total 24 TS while conventional rehabilitation program was given
  Interventions: Other: thermal stimulation
- thermal stimulation (innocuous) (Active Comparator): Heat:40-41°C and Cold:23-24°C alternately (intervention) 3 times /week and total 24 TS while conventional rehabilitation program was given
  Interventions: Other: thermal stimulation

INTERVENTIONS:
Other: thermal stimulation — hot and cold/warm and cool pads applying.
  Other Names: Thermal stimulation (FIRSTEK, Model-B401L,local company).

SUMMARY:
The thermal stimulation have been proven effective in upper extremity of stroke patients. Therefore, this study explored the efficacy of thermal stimulation in lower extremity of stroke patients.

DETAILED DESCRIPTION:
There are two groups of stroke patients (onset > 3 months) in this study. The independent factor is temperature of the alternated heat and cold applying.

ELIGIBILITY:
The inclusive criteria:

* first-ever stroke
* stroke onset > 3 months and < 3 years before the study enrollment
* unilateral hemiplegia
* ability to sit on a chair > 30 minutes independently
* able to follow verbal instructions
* age between 18 y/o and 80 y/o
* be willing to participate in this study and gave their informed consent

The exclusive criteria:

* skin disease, skin injuries, burns, or fresh scars over the TS application area
* contraindication of ice or heat application
* speech disorder or global aphasia
* musculoskeletal or cardiac disorders that could potentially interfere
* diabetic history or sensory impairment attributable to neuropathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The change score from baseline to post-treatment and baseline to 1M follow-up in the lower-limb subscale of the Stroke Rehabilitation Assessment of Movement(LE-STREAM) | pre, post, 1M follow-up
  The lower-limb subscale of the Stroke Rehabilitation Assessment of Movement (LE-STREAM) was assessed at the time before the first intervention (pre-assessment), the time after the 24th TS (post-assessment). The whole intervention was finished within 10 weeks. The third assessment was at 1M follow-up.
The change score from baseline to post-treatment and baseline to 1M follow-up in the mobility subscale of the Stroke Rehabilitation Assessment of Movement STREAM (Mob-STREAM) | pre, post, 1M follow-up
  The mobility subscale of the Stroke Rehabilitation Assessment of Movement STREAM (Mob-STREAM) was assessed at the time before the first intervention (pre-assessment), the time after the 24th TS (post-assessment). The whole intervention was finished within 10 weeks. The third assessment was at 1M follow-up.
The change score from baseline to post-treatment and baseline to 1M follow-up in the Functional Ambulation Category (FAC) | pre, post, 1M follow-up
  Functional Ambulation Category (FAC) was assessed at the time before the first intervention (pre-assessment), the time after the 24th TS (post-assessment). The whole intervention was finished within 10 weeks. The third assessment was at 1M follow-up.
The change score from baseline to post-treatment and baseline to 1M follow-up in the Barthel Index | pre, post, 1M follow-up
  Barthel Index (BI) was assessed at the time before the first intervention (pre-assessment), the time after the 24th TS (post-assessment). The whole intervention was finished within 10 weeks. The third assessment was at 1M follow-up.

SECONDARY OUTCOMES:
The change score from baseline to post-treatment and baseline to 1M follow-up in the Postural Assessment Scale for Stroke Patients (PASS) | pre, post, 1M follow-up
  Postural Assessment Scale for Stroke Patients (PASS) was assessed at the time before the first intervention (pre-assessment), the time after the 24th TS (post-assessment). The whole intervention was finished within 10 weeks. The third assessment was at 1M follow-up.
The change score from baseline to post-treatment and baseline to 1M follow-up in the Modified Ashworth Scale | pre, post, 1M follow-up
  Modified Ashworth Scale (MAS) was assessed at the time before the first intervention (pre-assessment), the time after the 24th TS (post-assessment). The whole intervention was finished within 10 weeks. The third assessment was at 1M follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Wen Hsin, graduated, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan, Taiwan